CLINICAL TRIAL: NCT04407065
Title: Double Trigger in Patients With Low Number of Oocytes Retrieved Per Number of Preovulatory Follicles. A Randomized Controlled Trial
Brief Title: Double Trigger in Patients With Low Number of Oocytes Retrieved Per Number of Preovulatory Follicles
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riyadh Fertility and Reproductive Health center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Double trigger/more oocytes
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Infertility, Female
Keywords: IVF; HCG; GnRH agonist trigger
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double trigger (Experimental): GnRH-agonist and HCG are used to trigger ovulation
  Interventions: Drug: Double trigger
- HCG (Active Comparator): HCG is used to trigger ovulation
  Interventions: Drug: HCG trigger

INTERVENTIONS:
Drug: Double trigger — Final follicular maturation is triggered by the co-administration of GnRH-agonist (Triptorelin acetate, decapeptyl 0.2 mg, Slough, United Kingdom) and 10000 IU of HCG, 40 and 34 h prior to oocyte retrieval, respectively
  Arms: Double trigger
Drug: HCG trigger — Final follicular maturation is triggered by a dose of 10000 IU of HCG 36 h prior to oocyte retrieval
  Arms: HCG

SUMMARY:
The aim of this randomized controlled trial is to determine whether co-administration of GnRH agonist and hCG for final oocyte maturation ( 40 and 34 h prior to oocyte retrieval , respectively) can increase the oocytes yield in patients with history of poor oocytes yield, despite normal response to COH, due to low (<50%) number of oocytes retrieved per number of follicles > 14 mm in diameter on day of hCG administration

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of poor oocytes yield in previous IVF attempt, despite normal response to COH, due to low (<50%) number of oocytes retrieved per number of follicles > 14 mm in diameter on day of hCG administration
* Patients with 6 to 15 mature follicles on the day oocyte trigger in the current IVF-ET attempt

Exclusion Criteria:

* Endometriosis
* PCOS

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 56 (Estimated)
Dates: Start 2020-05-30 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-02-02 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes retrieved | First day after oocyte retrieval

SECONDARY OUTCOMES:
clinical pregnancy rate | First 5 weeks after oocyte retrieval
  The presence of gestational sac detected by ultrasound examination

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, Prof., Study Director — Riyadh Fertility and Reproductive Health center
Locations (1):
- Riyadh Fertility and Reproductive Health center, Giza, Egypt

REFERENCES:
- [Background] Haas J, Zilberberg E, Dar S, Kedem A, Machtinger R, Orvieto R. Co-administration of GnRH-agonist and hCG for final oocyte maturation (double trigger) in patients with low number of oocytes retrieved per number of preovulatory follicles--a preliminary report. J Ovarian Res. 2014 Aug 2;7:77. doi: 10.1186/1757-2215-7-77. PMID 25296696